CLINICAL TRIAL: NCT02481440
Title: Repeated Subarachnoid Administrations of Human Umbilical Cord Mesenchymal Stem Cells in Treating Spinal Cord Injury
Brief Title: Repeated Subarachnoid Administrations of hUC-MSCs in Treating SCI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Limin Rong (Other)
Responsible Party: Sponsor-Investigator, Limin Rong, Director of Spine Surgery Department, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hUC-MSC-SCI
Record Dates: First submitted 2015-06-15; First posted 2015-06-25 (Estimated); Results first posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Spinal Cord Injuries
Keywords: human umbilical cord mesenchymal stem cells; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hUC-MSC Transplantation (Experimental): Repeated intrathecal administrations of 1x10E6 human umbilical cord mesenchymal stem cells per kg in subjects with spinal cord injury with an interval of one month between each administration
  Interventions: Biological: human umbilical cord mesenchymal stem cells (hUC-MSCs)

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cells (hUC-MSCs) — Four times of intrathecal administrations of hUC-MSCs
  Other Names: umbilical cord mesenchymal stem cells

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of repeated intrathecal administrations of allogeneic human umbilical cord mesenchymal stem cells for the treatment of spinal cord injury.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a devastating disease and often leads to lifelong disability, muscle spasm, sensory deficits, autonomic disturbances, as well as bowel and bladder incontinence, all of which can cause tremendous troubles to patients but are lack of any effective treatment up to now. SCI is not only a severe healthy problem but also a great social burden. To the best of our knowledge, cell therapy seems to be a promising alternative for the treatment of SCI due to numerous advantages. However, cytotherapy is still in its infancy since there are many disparities and uncertainties regarding subject selection, cellular type, transplantation timing, administration dose and deliver route in clinical trial protocols. Hence, a standardized well-designed clinical study is urgently required for the safe and effective treatment of SCI.

In this study, complete or incomplete cervical, thoracic, and thoracolumbar SCI subjects were recruited to join in a prospective, single-center, single-arm clinical trial. Intervention is four times of subarachnoid administration of allogeneic hUC-MSCs. During the intervention and follow-up periods of this trial, any adverse event was identified rapidly and managed properly. The maximum intensity and relationship of any adverse event with hUC-MSCs administration were identified.The primary efficacy indicator is American spinal injury association (ASIA) total score at the fourth follow-up and SCI Functional Rating Scale of the International Association of Neurorestoratology (IANR-SCIFRS) total score at the fourth follow-up. Secondary efficacy indicators are these two indicators at the remaining time points, scores of pin prick, light touch, motor and sphincter, muscle spasticity and spasm, autonomic system, bladder and bowel functions, residual urine volume. Subgroup analysis of primary efficacy indicators was also performed.

In this trial, informed consent forms that had the approval of the institutional review board were obtained from all participants before recruitment. In this clinical study, subarachnoid transplantation of hUC-MSCs was performed a total of four times per subject with the delivery dose of 1×10E6 cells/kg. After the completion of cytotherapy, subject was regularly followed up in the hospital at four time points, determined at 1, 3, 6, and 12 months following the final administration of hUC-MSCs. At each time point of administration (the first, second, third, and fourth transplantation) and follow-up (the first, second, third, and fourth follow-up), safety and efficacy indicators were collected accordingly by two independent assessors.

ELIGIBILITY:
Inclusion Criteria:

1. complete or incomplete trauma-induced SCI [American Spinal Injury Association (ASIA) Impairment Scale classification: A-D] that happened at least two months before recruitment;
2. aged between 18 and 65 years;
3. agreed to participate in this study voluntarily and be regularly followed up for 12 months after the completion of hUC-MSCs administration

Exclusion Criteria:

1. ankylosing spondylitis, myelitis, or vascular abnormalities within the spinal cord parenchyma;
2. severe comorbidities, including but not limited to craniocerebral injury, cutaneous back infection, psychiatric disease, or cancer;
3. pregnancy or lactation (for females);
4. predicted lifespan of less than 12 months following the end of hUC-MSCs transplantation;
5. participation in any other stem cell-related clinical trials that might affect accurate neurological evaluations in the present trial;
6. any medical condition that, in the opinion of investigators, may pose a safety risk to any subject in this study, confound safety or efficacy assessments, or interfere with study participation

Rejection Criteria:

1. misdiagnosis;
2. use of any medication that may significantly impact the assessment accuracy of stem cell engraftment;
3. absence of any evaluation outcome at any time point during the follow-up period

Cessation Criteria:

1. individual wishes of the subjects;
2. occurrence of any stem cell-associated serious adverse event (SAE) that may aggravate neurological dysfunction, or require prolongation of existing hospitalization, or need hospital readmission, or impair consciousness, or be life-threatening, or even lead to death in any subject;
3. detection of any major mistake in the present protocol during the implementation of this clinical trial;
4. the national administration agency requires the clinical trial to be halted

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min Li Rong, M.D., Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- hUC-MSC Transplantation: Four times of intrathecal administrations of 1x10E6 human umbilical cord mesenchymal stem cells per kg in subjects with spinal cord injury with an interval of one month between each administration
Period: Overall Study
Arm/Group | hUC-MSC Transplantation
Started | 102
Completed | 41
Not Completed | 61

BASELINE CHARACTERISTICS:
Arm/Group | hUC-MSC Transplantation
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 41
Chronicity of SCI [Mean (Standard Deviation); unit: months] | 45.15 (59.78)

OUTCOME MEASURES:

1. Primary Outcome: American Spinal Injury Association (ASIA) Total Score at the Fourth Follow-up
Description: American Spinal Injury Association (ASIA) form is used to assess ASIA total score (Range: 0-324 scores). The higher scores mean a better outcome.
Time Frame: at 12 months following the final administration of hUC-MSCs
Measure: Mean (Standard Deviation); unit: score
Arm/Group | hUC-MSC Transplantation
Number analyzed (Participants) | 41
score | 183.88 (69.76)

2. Primary Outcome: SCI Functional Rating Scale of the International Association of Neurorestoratology (IANR-SCIFRS) Total Score at the Fourth Follow-up
Description: SCI Functional Rating Scale of the International Association of Neurorestoratology (IANR-SCIFRS) form is used to assess IANR-SCIFRS total score (Range: 0-51 scores). The higher scores mean a better outcome.
Time Frame: at 12 months following the final administration of hUC-MSCs
Measure: Mean (Standard Deviation); unit: score
Arm/Group | hUC-MSC Transplantation
Number analyzed (Participants) | 41
score | 29.49 (10.47)

3. Secondary Outcome: American Spinal Injury Association (ASIA) Total Score
Description: as for outcome 1
Time Frame: at first, second, third, and fourth transplantation and 1, 3, 6 months following the final administration of hUC-MSCs
Measure: Mean (Standard Deviation); unit: score
Arm/Group | hUC-MSC Transplantation
Number analyzed (Participants) | 41
score
  3rd follow-up | 182.44 (71.00)
  2nd follow-up | 178.39 (71.51)
  1st follow-up | 176.05 (71.88)
  4th transplantation | 172.00 (73.51)
  3rd transplantation | 168.41 (74.16)
  2nd transplantation | 163.80 (72.53)
  1st transplantation | 158.15 (70.93)

4. Secondary Outcome: SCI Functional Rating Scale of the International Association of Neurorestoratology (IANR-SCIFRS) Total Score
Description: as for outcome 2
Time Frame: at first, second, third, and fourth transplantation and 1, 3, 6 months following the final administration of hUC-MSCs
Measure: Mean (Standard Deviation); unit: score
Arm/Group | hUC-MSC Transplantation
Number analyzed (Participants) | 41
score
  3rd follow-up | 28.93 (10.26)
  2nd follow-up | 28.44 (10.28)
  1st follow-up | 27.56 (10.03)
  4th transplantation | 26.85 (10.36)
  3rd transplantation | 26.05 (10.15)
  2nd transplantation | 25.71 (10.32)
  1st transplantation | 24.54 (9.82)

5. Secondary Outcome: International Standards to Document Remaining Autonomic Function After Spinal Cord Injury (ISAFSCI) Score
Description: International Standards to document remaining Autonomic Function after Spinal Cord Injury (ISAFSCI) form is used to assess ISAFSCI score (autonomic nervous function) (Range: 5-32 scores). The higher scores mean a better outcome.
Time Frame: at first transplantation and 12 months following the final administration of hUC-MSCs
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | hUC-MSC Transplantation
Number analyzed (Participants) | 41
score
  4th follow-up | 12 [11 to 14]
  1st transplantation | 11 [10 to 12]

6. Secondary Outcome: Penn Scale
Description: Penn scale form is used to assess muscle spasm (Range: 0-4 scores). The higher scores mean a worse outcome.
Time Frame: at first transplantation and 12 months following the final administration of hUC-MSCs
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | hUC-MSC Transplantation
Number analyzed (Participants) | 41
score
  4th follow-up | 1 [0 to 2]
  1st transplantation | 1 [0 to 3]

7. Secondary Outcome: Modified Ashworth Scale
Description: Modified Ashworth scale form is used to assess muscle spasticity (Range: 0-16 scores). The higher scores mean a worse outcome.
Time Frame: at first transplantation and 1, 3, 12 months following the final administration of hUC-MSCs
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | hUC-MSC Transplantation
Number analyzed (Participants) | 41
score
  4th follow-up | 2 [0 to 4]
  2nd follow-up | 2 [0 to 4]
  1st follow-up | 2.5 [0 to 4.5]
  1st transplantation | 3 [0 to 6]

8. Secondary Outcome: Geffner Scale
Description: Geffner scale form is used to assess bladder function (Range: 0-7 scores). The higher scores mean a better outcome.
Time Frame: at first transplantation and 12 months following the final administration of hUC-MSCs
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | hUC-MSC Transplantation
Number analyzed (Participants) | 41
score
  4th follow-up | 3 [2 to 4]
  1st transplantation | 2 [0 to 4]

9. Secondary Outcome: Neurogenic Bowel Dysfunction (NBD) Scale
Description: Neurogenic Bowel Dysfunction (NBD) scale form is used to assess bowel function (Range: 0-47 scores). The higher scores mean a worse outcome.
Time Frame: at first transplantation and 12 months following the final administration of hUC-MSCs
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | hUC-MSC Transplantation
Number analyzed (Participants) | 41
score
  4th follow-up | 3 [2 to 10]
  1st transplantation | 6 [2 to 12.5]

10. Secondary Outcome: Residual Urine Volume
Description: Ultrasonic examination is used to assess residual urine volume
Time Frame: at first transplantation and 12 months following the final administration of hUC-MSCs
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | hUC-MSC Transplantation
Number analyzed (Participants) | 41
ml
  4th follow-up | 27.90 [8.83 to 88.50]
  1st transplantation | 67.65 [31.58 to 144.50]

ADVERSE EVENTS:
Time Frame: During the intervention and follow-up periods of this trial, up to 16 months, any AE was identified and collected.
Arm/Group | hUC-MSC Transplantation
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 44/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hUC-MSC Transplantation (N=102)
transient increase of muscle tension (Nervous system disorders) | 2 (6)
fever (Immune system disorders) | 25 (54)
headache (Nervous system disorders) | 14 (16)
dizziness (Nervous system disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT02481440/Prot_SAP_000.pdf